CLINICAL TRIAL: NCT02814799
Title: Study of the Effects of the Bone Tissue on the Generation of Thrombine
Brief Title: Effects of the Bone Tissue on the Haemostasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PJ12077
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Dental Disease
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- bone donors
  Interventions: Other: bone removal

INTERVENTIONS:
Other: bone removal

SUMMARY:
The research for a haemostasis and for an effective osseous healing are a major stake in oral surgery. The use of glues of fibrin, amplifying the polymerization of the fibrin during the haemostasis is known to reduce the risk of post-operative bruise and accelerate the healing but these glues present the inconvenience to be by-products of the blood, not devoid of infectious risk.

DETAILED DESCRIPTION:
Thrombinography is a functional exploration of the haemostasis allowing the characterization of the kinetics and the amount of thrombin. Its principle bases on the recording of the activity of the in vitro thrombin, by fluorometry. The formed thrombin leads a signal by activation of the fluorogenic substrates. The intensity of the received signal is correlated in the generation of thrombin by comparative measure of the fluorescence of a standard sample of thrombinic activity known. The analysis is realized by a specific software: Thrombinoscope®. The used reactional environment is a poor Plasma in platelet (PPP).

The software defines the quantity of thrombin generated (nM) according to time (in minute) and calculate the values of:

* Lag time: latent period before the beginning of synthesis of thrombin.
* Start Tail: duration of the process.
* Peak: peak of thrombin, is the maximal rate of generated thrombin.
* ETP (Endogenous Thrombin Potential): area under the curve representing the total potential of generation of thrombin.
* Time to Peak: time required to reach the peak of thrombin. It is these values which will serve as criteria of evaluation for our study.

Osseous type

The cancellous bone is majority in the short bones and the epiphyses of the long bones. It is crisp, constituted by fine osseous patches arranged in a not concentric way around wide open cavities, filled with bone marrow rich in cells, and richly vascularized. The cancellous bone is surrounded with compact bone. At the level of tooth sockets, this osseous type is found in particular at the level of interradicular septa.

The compact bone establishes the cortical. It is dense, consisted of systems of Havers. Every system is formed by a reduced central channel containing some vascularized connective tissue, and thick, concentric osseous small strips, in and between which prepares ostéocytes. This osseous type is situated at the alveolar level in the external part.

Inhibitors

To verify the possible ways involved in the thrombin formation, the investigators shall use specific inhibitors of these likely ways of activation:

* An inhibitor of the extrinsic way of the coagulation: an antibody anti tissue factor.
* An inhibitor of the intrinsic way of the coagulation: the bovine aprotinin.
* An inhibitor of phospholipids: the annexin V. Methodology of the Research

Plan of investigation

* Information of the eligible patients for the study (patients requiring dental extractions with bone removal) concerning the methods and the objectives of the research by means of the information note.
* If the patient agrees to participate in the study, realization of osseous takings and conditioning of the osseous takings for freezing in the liquid nitrogen.
* Put in touch by the osseous takings with some plasma (from pools of plasma used in laboratory for the calibration of the various automatous) and measure of the genesis of thrombin by thrombinography.

To make this measure, the osseous fragments will be put down at the bottom of the wells of the microplate then 10µL of buffer HBS will be added. The fragmentation of the osseous takings will be realized by means of a sterile material and by limiting the time of manipulation except environment.

Every sample will be handled triplicate there. Two wells will be dedicated to the standard thrombin (20µL). Two controls will be used: - positive control: 10µL of tissue factor, in the concentration of 1 or 5 pM and 10µL of PPL in the dilution of 1/100 will be used.

- Negative control: 20µL of physiological salt solution will be used. Eighty microliters of plasma are going to be put down in each of the wells. Fifty microliters of fluorescent substratum will be added to the mixture buffer - substratum fluorogenic beforehand prepared and the device is going to distribute 20µL some mixture in each of the wells, thus containing in the end 120µL.

The measures were made every 20 seconds during 60 minutes by the Fluoroskan Ascent Reader. The Thrombinoscope softwar® (Version 3.0.0.29, Maastricht) converts the intensity of fluorescence nM of thrombin according to the time.

The results of the measures will be grouped in cancellous bone, compact bone, control FT1pM, control FT5pM and secondarily averaged.

According to the obtained results, samples (compact and\or cancellous) positive for the genesis of thrombin will be analyzed in the presence of specific inhibitors of the various possible ways of activation of the coagulation. Calibrations will be made to choose the most appropriate concentration in inhibitors.

Logistics of the study

An information concerning the objectives and the modalities of the study will be given to every patient benefiting from one or several dental extractions with bone removal. If the patient agrees to participate in the study (oral agreement), the osseous taking, associated automatically with the dental extraction will be kept.

After taking, the osseous fragments will be immersed in a solution of cryopreservation beforehand prepared, then put down in a freezer in -70°C during a minimum of 24 hours before being immersed in the liquid nitrogen.

The measures of trhombinography will be realized at the rate of an analysis every other week, adaptable periodicity according to the number of recruitment made during the period.

ELIGIBILITY:
Inclusions criteria

Will be included in this study:

* The patients requiring dental extractions with bone removal
* The patients agreeing to participate in the search

Exclusions criteria

Will not be included in this study:

* Minor patients.
* Patients protected by the law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusive patients will be all the patients requiring dental extractions with bone removal, taken care in the department of odontology of the CHU of Reims and agreeing to participate in the study. Only these patients form the group of observed patients. The duration of participation of the patient in the study is punctual, the time of the osseous taking.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
thrombin quantification | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France